CLINICAL TRIAL: NCT01809210
Title: A Phase I, Open Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Selumetinib (AZD6244; ARRY-142886) in Combination With First Line Chemotherapy Regimens in Patients With Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Assess Safety & Efficacy of Selumetinib When Given in Combination With Standard First Line Treatment for Advanced Non-small Cell Lung Cancer
Acronym: SELECT-3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1532C00070; EudraCT number: 2012-005202-22
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Locally Advanced or Metastatic NSCL Cancer Stage IIIB IV
Keywords: MEK1/2 inhibitor,; Non Small Cell Lung Cancer,; metastatic,; first line treatment for Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasm Metastasis | interventions — AZD 6244; Gemcitabine; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Selumetinib+standard chemotherapy (Experimental): Selumetinib plus gemcitabine; or pemetrexed and cisplatin or carboplatin
  Interventions: Drug: selumetinib; Drug: gemcitabine; Drug: cisplatin; Drug: carboplatin; Drug: pemetrexed

INTERVENTIONS:
Drug: selumetinib — 2 x 25mg capsules bd continuously in cohort 1 (with gemcitabine and cisplatin). If tolerated - next cohort 3 x 25mg capsules bd continuously. if higher doses are explored, required number of capsules will be provided. Option to administer on D2-19 of each 21 day cycle if required to assess tolerability of combinations with chemotherapy
Drug: gemcitabine — 1250 mg/m2 iv on Day 1 and 8 of each 21 day cycle. If combination not tolerated, option to give 1000 mg/m2 iv on Day 1 and Day 8 of each 21 day cycle
Drug: cisplatin — 75 mg/m2 iv on Day 1 of each 21 day cycle. If combination not tolerated, option to give 50 mg/m2 iv on Day 1 or 25mg/m2 iv on Day 1 and Day 8 of each 21 day cycle
Drug: carboplatin — If it is not possible to identify a tolerable combination of selumetinib, gemcitabine and cisplatin, cisplatin may be replaced with carboplatin (AUC5) iv on Day 1 of each 21 day cycle
Drug: pemetrexed — Gemcitabine may be replaced with pemetrexed 500 mg/m2 iv on Day 1 of each 21 day cycle.

SUMMARY:
This is a Phase I, open label multicentre study of selumetinib administered orally in combination with first line chemotherapy regimens to patients with advanced/metastatic NSCLC. The study has been designed to allow an investigation of the optimal dose of selumetinib in combination with various standard first line double-platinum chemotherapy regimens. Initial assessment will be based on tolerability of selumetinib in combination with one or more selected regimens that are considered to be tolerated also being assessed for preliminary evidence of activity.

This study is a dose finding and optional cohort expansion; In addition all patients will be assessed for anti-cancer efficacy of the combination of selumetinib and chemotherapy.

DETAILED DESCRIPTION:
A Phase I, Open Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Selumetinib (AZD6244; ARRY-142886) in Combination with First Line Chemotherapy Regimens in Patients with Non-Small Cell Lung Cancer (NSCLC)

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed, written and dated consent prior to any study specific procedures
* Male or female, aged 18 years or older
* Histological or cytological confirmation of locally advanced or metastatic NSCLC (IIIB-IV)
* Female patients must not be breast-feeding and have a negative pregnancy test prior to start of dosing or must have evidence of non-child-bearing potential
* Patients must be eligible to receive treatment with the platinum doublet combination with which selumetinib is being combined and in accordance with the local product information

Exclusion Criteria:

* Prior chemotherapy or other systemic anti-cancer treatment for advanced NSCLC.
* Prior surgery or radiotherapy within 6 months or palliative radiotherapy within 4 weeks of start of study treatment.
* Female patients who are breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
* Another primary malignancy within 5 years of starting study treatment, except for adequately treated basal or squamous cell carcinoma of the skin or cancer of the cervix in situ.
* As judged by the Investigator, any evidence of severe or uncontrolled systemic diseases, active bleeding diatheses, renal transplant, or active infection

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-04-04 (Actual); Primary Completion 2016-01-04 (Actual); Study Completion 2016-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella Mariani, MD, Study Director — AstraZeneca UK, MSD; Emma Dean, BMEDSCI, BM, BS, PHD, Principal Investigator — The Christie NHS Foundation Trust, UK; Fiona Blackhall, PhD, FRCP, Principal Investigator — The Christie NHS Foundation Trust Clinical Trials Unit; UK
Locations (4):
- United Kingdom (4):
  - Research Site, Glasgow
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Newcastle upon Tyne

REFERENCES:
- See also: D1532C00070revisedCSP-2_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1179&filename=D1532C00070revisedCSP-2_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled into dose-finding cohorts to evaluate escalating doses of selumetinib (AZD6244; ARRY-142886) to determine the maximum tolerated dose in combination with standard first-line chemotherapy regimens. Chemotherapy was administered on Day 1 (and Day 8 for gemcitabine) of each 3-week cycle.
Pre-assignment Details: Data cut off (DCO) was 7 Jan 16. DCO was defined as the earliest of 12 (±1) weeks after last patient started, or 28 days after final patient discontinued, selumetinib or chemotherapy doublet regimen.
Groups:
- Cohort 1 sel50, Gem, Cis: selumetinib 50mg bd, gemcitabine 1250mg/m2 , cisplatin 75mg/m2
- Cohort 2 sel50, Gem, Carb: selumetinib 50mg bd, gemcitabine 1250mg/m2 , carboplatin 5 units
- Cohort 3 sel75, Gem, Cis: selumetinib 75mg bd, gemcitabine 1250mg/m2 , cisplatin 75mg/m2
- Cohort 4 sel150, Pem, Carb: selumetinib 50mg bd, pemetrexed 500 mg/m2, carboplatin 5 units
- Cohort 5 sel75, Pem, Carb: selumetinib 75mg bd, pemetrexed 500 mg/m2, carboplatin 5 units
- Cohort 6 sel75, Pem, Cis: selumetinib 75mg bd, pemetrexed 500 mg/m2, cisplatin 75mg/m2
- Cohort 7 sel100, Pem, Carb: selumetinib 100mg bd, pemetrexed 500 mg/m2, carboplatin 5 units
Period: Overall Study
Arm/Group | Cohort 1 sel50, Gem, Cis | Cohort 2 sel50, Gem, Carb | Cohort 3 sel75, Gem, Cis | Cohort 4 sel150, Pem, Carb | Cohort 5 sel75, Pem, Carb | Cohort 6 sel75, Pem, Cis | Cohort 7 sel100, Pem, Carb
Started | 3 | 9 | 7 | 3 | 6 | 15 | 12
Completed | 2 | 8 | 4 | 2 | 4 | 12 | 7
Not Completed | 1 | 1 | 3 | 1 | 2 | 3 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 1 | 0 | 4
Not completed — Death | 1 | 1 | 2 | 0 | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 sel50, Gem, Cis | Cohort 2 sel50, Gem, Carb | Cohort 3 sel75, Gem, Cis | Cohort 4 sel150, Pem, Carb | Cohort 5 sel75, Pem, Carb | Cohort 6 sel75, Pem, Cis | Cohort 7 sel100, Pem, Carb | Total
Number analyzed (Participants) | 3 | 9 | 7 | 3 | 6 | 15 | 12 | 55
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.7 (3.79) [56 to 63] | 69.2 (3.53) [65 to 76] | 55.1 (8.65) [39 to 65] | 64.7 (7.23) [60 to 73] | 59.5 (5.28) [54 to 66] | 61.8 (5.86) [54 to 71] | 60.2 (8.39) [46 to 73] | 61.5 (7.45) [39 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 3 | 1 | 4 | 5 | 7 | 26
  Male | 2 | 4 | 4 | 2 | 2 | 10 | 5 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Or African American | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3
  Other | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  White | 2 | 9 | 7 | 3 | 5 | 13 | 11 | 50

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT) Events in Chemotherapy in Combination With Selumetinib
Description: Any toxicity not attributable to the disease or disease-related processess under investigation, considered related to the combination of chemotherapy plus selumetinib, which occurs within the timeframe and is dose limiting
Time Frame: The first dose on Cycle 1 Day 1 up to the time before dosing on Cycle 2 Day 1, assessed up to 3 weeks
Population: Safety analysis set - all patients who received at least 1 dose of selumetinib.
Measure: Number; unit: participants
Arm/Group | Cohort 1 sel50, Gem, Cis | Cohort 2 sel50, Gem, Carb | Cohort 3 sel75, Gem, Cis | Cohort 4 sel150, Pem, Carb | Cohort 5 sel75, Pem, Carb | Cohort 6 sel75, Pem, Cis | Cohort 7 sel100, Pem, Carb
Number analyzed (Participants) | 3 | 9 | 7 | 3 | 6 | 15 | 12
participants
  Evaluable patients | 3 | 7 | 4 | 3 | 6 | 12 | 6
  Evaluable patients with a DLT Event | 0 | 2 | 1 | 0 | 0 | 1 | 1

2. Secondary Outcome: Best Objective Response
Description: The best response a patient has had during their time in the study up until RECIST progression or last valuable assessment in the absence of RECIST progression. Per Response Evaluation Criteria In Solid Tumours (RECIST version 1.1) for target lesions (TL) and assessed by MRI or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progressive Disease (PD); Progressive Disease (PD), >=20% increase in the sum of the longest diameter of target lesions, the sum must also demonstrate an absolute increase of >=5mm; Complete Response (CR), disappearance of all target lesions, any pathological lymph nodes selected as TLs must have a reduction in short axis to <10mm
Time Frame: Screening, week 6 and week 12
Population: Tumour response analysis set - dosed patients with a baseline tumour assessment.
Measure: Number; unit: participants
Arm/Group | Cohort 1 sel50, Gem, Cis | Cohort 2 sel50, Gem, Carb | Cohort 3 sel75, Gem, Cis | Cohort 4 sel150, Pem, Carb | Cohort 5 sel75, Pem, Carb | Cohort 6 sel75, Pem, Cis | Cohort 7 sel100, Pem, Carb
Number analyzed (Participants) | 3 | 9 | 7 | 3 | 6 | 15 | 12
participants
  Complete response | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial response | 1 | 2 | 2 | 1 | 1 | 2 | 2
  Unconfirmed complete or partial response | 0 | 3 | 0 | 0 | 2 | 2 | 2
  Stable disease | 0 | 1 | 2 | 2 | 3 | 7 | 6
  RECIST progression | 2 | 0 | 1 | 0 | 0 | 1 | 1
  Death | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Incomplete post-baseline assessments | 0 | 3 | 2 | 0 | 0 | 2 | 1

3. Secondary Outcome: Percentage Change From Baseline at 6 Weeks in Target Lesion Size
Description: The percentage change in the sum of the diameters of target lesions
Time Frame: Week 6
Population: Tumour response analysis set - dosed patients with a baseline tumour assessment.
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Cohort 1 sel50, Gem, Cis | Cohort 2 sel50, Gem, Carb | Cohort 3 sel75, Gem, Cis | Cohort 4 sel150, Pem, Carb | Cohort 5 sel75, Pem, Carb | Cohort 6 sel75, Pem, Cis | Cohort 7 sel100, Pem, Carb
Number analyzed (Participants) | 3 | 9 | 7 | 3 | 6 | 15 | 12
% change | -7.5 (19.79) | -29.3 (11.15) | -10.4 (24.45) | -14.7 (1.91) | -24.4 (32.60) | -18.9 (10.55) | -18.4 (19.58)

4. Secondary Outcome: Best Percentage Change From Baseline in Target Lesion Size
Description: The best percentage change in tumour size a patient has had during their time in the study up until RECIST progression or last valuable assessment in the absence of RECIST progression. Percentage change was derived at each visit by the percentage change in the sum of the diameters of target lesions
Time Frame: Screening, week 6 and week 12
Population: Tumour response analysis set - dosed patients with a baseline tumour assessment.
Measure: Mean (Standard Deviation); unit: % change
Arm/Group | Cohort 1 sel50, Gem, Cis | Cohort 2 sel50, Gem, Carb | Cohort 3 sel75, Gem, Cis | Cohort 4 sel150, Pem, Carb | Cohort 5 sel75, Pem, Carb | Cohort 6 sel75, Pem, Cis | Cohort 7 sel100, Pem, Carb
Number analyzed (Participants) | 3 | 9 | 7 | 3 | 6 | 15 | 12
% change | -11.9 (26.52) | -34.6 (8.11) | -41.3 (21.25) | -28.3 (15.25) | -34.7 (33.30) | -24.4 (14.71) | -25.4 (20.51)

5. Secondary Outcome: Objective Response Rate (ORR)
Description: The number of patients who had at least 1 confirmed visit response of Complete Response (CR) or Partial Response (PR) prior to any evidence of progression. Per Response Evaluation Criteria In Solid Tumours (RECIST version 1.1) for target lesions (TL) and assessed by MRI or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Complete Response (CR), disappearance of all target lesions, any pathological lymph nodes selected as TLs must have a reduction in short axis to <10mm; Objective Response Rate (ORR) = CR + PR
Time Frame: Up until progression or last evaluable assessment in the absence of progression, up to 9 months
Population: Tumour response analysis set - dosed patients with a baseline tumour assessment.
Measure: Number; unit: participants
Arm/Group | Cohort 1 sel50, Gem, Cis | Cohort 2 sel50, Gem, Carb | Cohort 3 sel75, Gem, Cis | Cohort 4 sel150, Pem, Carb | Cohort 5 sel75, Pem, Carb | Cohort 6 sel75, Pem, Cis | Cohort 7 sel100, Pem, Carb
Number analyzed (Participants) | 3 | 9 | 7 | 3 | 6 | 15 | 12
participants | 1 (26.52) | 2 (8.11) | 2 (21.25) | 1 (15.25) | 1 (33.30) | 2 (14.71) | 2 (20.51)

6. Secondary Outcome: AUC (0-tau)
Description: Area under the concentration time curve (AUC) over a dosing interval at steady state (0-tau)
Time Frame: Cycle 2 Day1, pre-dose, 0.5, 1, 1.5, 2, 4, 8, 10 hours post dose
Population: Pharmacokinetic analysis set - patients with sufficient samples to provide an adequate PK profile for determination of PK parameters with no important adverse events or protocol deviations that may have impacted PK
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Cohort 1 sel50, Gem, Cis | Cohort 2 sel50, Gem, Carb | Cohort 3 sel75, Gem, Cis | Cohort 4 sel150, Pem, Carb | Cohort 5 sel75, Pem, Carb | Cohort 6 sel75, Pem, Cis | Cohort 7 sel100, Pem, Carb
Number analyzed (Participants) | 3 | 9 | 7 | 3 | 6 | 15 | 12
h*ng/mL | NA (NA) — Not calculated as only 2 patients provided sufficient PK samples for AUC calculation and therefore geometric mean was not calculated. (Min 2130, Max 2240) | 3571 (42.13) | 3339 (15.08) | 4813 (30.93) | 4366 (48.14) | 4116 (33.92) | 5202 (52.94)

7. Secondary Outcome: Cmax,ss
Description: Maximum plasma concentration at steady state
Time Frame: Cycle 2 Day1, pre-dose, 0.5, 1, 1.5, 2, 4, 8, 10 hours post dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 sel50, Gem, Cis | Cohort 2 sel50, Gem, Carb | Cohort 3 sel75, Gem, Cis | Cohort 4 sel150, Pem, Carb | Cohort 5 sel75, Pem, Carb | Cohort 6 sel75, Pem, Cis | Cohort 7 sel100, Pem, Carb
Number analyzed (Participants) | 3 | 9 | 7 | 3 | 6 | 15 | 12
ng/mL | 476.7 (51.12) | 1222 (59.86) | 1487 (23.09) | 1615 (27.71) | 1375 (40.21) | 1364 (57.78) | 2309 (35.99)

8. Secondary Outcome: Tmax,ss
Description: Time to reach maximum plasma concentration at steady state
Time Frame: Cycle 2 Day1, pre-dose, 0.5, 1, 1.5, 2, 4, 8, 10 hours post dose
Population: as for outcome 6
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 sel50, Gem, Cis | Cohort 2 sel50, Gem, Carb | Cohort 3 sel75, Gem, Cis | Cohort 4 sel150, Pem, Carb | Cohort 5 sel75, Pem, Carb | Cohort 6 sel75, Pem, Cis | Cohort 7 sel100, Pem, Carb
Number analyzed (Participants) | 3 | 9 | 7 | 3 | 6 | 15 | 12
h | 1.00 (51.12) [1.00 to 1.60] | 1.25 (23.09) [1.00 to 1.50] | 1.00 (57.78) [0.58 to 1.00] | 1.00 (59.86) [1.00 to 1.50] | 1.75 (27.71) [0.50 to 2.03] | 1.48 (40.21) [0.50 to 2.75] | 1.50 (35.99) [1.00 to 2.00]

9. Secondary Outcome: CL/F
Description: Apparent oral plasma clearance
Time Frame: Cycle 2 Day1, pre-dose, 0.5, 1, 1.5, 2, 4, 8, 10 hours post dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort 1 sel50, Gem, Cis | Cohort 2 sel50, Gem, Carb | Cohort 3 sel75, Gem, Cis | Cohort 4 sel150, Pem, Carb | Cohort 5 sel75, Pem, Carb | Cohort 6 sel75, Pem, Cis | Cohort 7 sel100, Pem, Carb
Number analyzed (Participants) | 3 | 9 | 7 | 3 | 6 | 15 | 12
L/h | NA (NA) — Not calculated as only 2 patients provided sufficient PK samples for CL/F calculation and therefore geometric mean was not calculated. (Min 22.3, Max 23.5) | 14.72 (5.156) | 22.64 (3.521) | 10.72 (3.328) | 18.82 (9.777) | 19.08 (5.881) | 21.02 (9.857)

ADVERSE EVENTS:
Time Frame: Adverse Events are collected throughout the study, from informed consent until the end of follow-up, which is defined as 28 +/- 7 days after selumetinib is discontinued. Patients were expected to receive up to 6 cycles (18 wks) of chemotherapy.
Arm/Group | Cohort 1 sel50, Gem, Cis | Cohort 2 sel50, Gem, Carb | Cohort 3 sel75, Gem, Cis | Cohort 4 sel150, Pem, Carb | Cohort 5 sel75, Pem, Carb | Cohort 6 sel75, Pem, Cis | Cohort 7 sel100, Pem, Carb
Serious Adverse Events (participants affected / at risk) | 1/3 | 6/9 | 3/7 | 2/3 | 3/6 | 9/15 | 9/12
Other Adverse Events (participants affected / at risk) | 3/3 | 9/9 | 7/7 | 3/3 | 6/6 | 15/15 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 sel50, Gem, Cis (N=3) | Cohort 2 sel50, Gem, Carb (N=9) | Cohort 3 sel75, Gem, Cis (N=7) | Cohort 4 sel150, Pem, Carb (N=3) | Cohort 5 sel75, Pem, Carb (N=6) | Cohort 6 sel75, Pem, Cis (N=15) | Cohort 7 sel100, Pem, Carb (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Retinal vein occlusion (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mediastinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 sel50, Gem, Cis (N=3) | Cohort 2 sel50, Gem, Carb (N=9) | Cohort 3 sel75, Gem, Cis (N=7) | Cohort 4 sel150, Pem, Carb (N=3) | Cohort 5 sel75, Pem, Carb (N=6) | Cohort 6 sel75, Pem, Cis (N=15) | Cohort 7 sel100, Pem, Carb (N=12)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 5 (7) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (9) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 6 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Conjunctival oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 6 (6)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (6) | 4 (5) | 2 (2) | 2 (2) | 6 (7) | 9 (13)
Diarrhoea (Gastrointestinal disorders) | 2 (4) | 5 (21) | 4 (7) | 1 (2) | 3 (8) | 9 (16) | 6 (8)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 3 (5)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (9) | 5 (13) | 5 (22) | 3 (4) | 5 (8) | 8 (15) | 10 (14)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retching (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 3 (5) | 1 (1) | 1 (1) | 3 (4) | 2 (3)
Tongue ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (8) | 4 (8) | 4 (19) | 1 (1) | 4 (9) | 6 (12) | 7 (13)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fat tissue increased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (3) | 6 (8) | 3 (4) | 1 (1) | 2 (2) | 9 (13) | 7 (11)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 4 (5)
Peripheral swelling (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angular cheilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 3 (4)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Abnormal weight gain (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 4 (4) | 2 (5) | 0 (0) | 3 (3) | 4 (4) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ketosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aphonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 5 (5)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2) | 3 (6) | 1 (3) | 2 (2) | 5 (6) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perineal fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perineal ulceration (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 2 (2) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5) | 0 (0) | 1 (1) | 3 (4) | 1 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plantar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 5 (5) | 2 (2) | 1 (2) | 8 (10) | 6 (6)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (4)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No